CLINICAL TRIAL: NCT04517136
Title: Impact of Perceived Control on Operational Strain: a Study of COVID-19 Pandemic Caregivers and Military Personnel on Operational Missions
Acronym: COVID-TRUST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-28; 2020-A01937-32 (Other: IDRCB)
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Covid19; SARS-CoV Infection; Burnout, Caregiver; Burnout, Professional
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Caregiver Burden; Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assessment of work-related stress — Assessment of burnout, mindfulness, interoceptive awareness, anxiety, post-traumatic stress disorder, coping flexibility and sleep through questionnaires.
Biological: Saliva sample collection — Saliva sample is collected before and after emotional stimulation in order to measure resting-state allostatic load biomarkers: Dehydroepiandrosterone (DHEA), cortisol and chromogranin A levels
Device: Cardiac and electrodermal recordings — Electrocardiogram and electrodermal activity (tonic and phasic) is collected at rest and after emotional stimulation.
Behavioral: Assessment of behavioral response to emotional stimulation — Emotional stimulation involves asking the participants to remember a recent event related to the COVID-19 crisis that has been emotionally difficult for them.
  Perceived stress, situational awareness and emotions is assessed after emotional stimulation through questionnaires.

SUMMARY:
Stress is underpinned by a biological reaction of the organism allowing the production of energy to respond to a change in the environment (or stressor). Stress reaction is expressed in behavioural, cognitive, emotional and physiological terms. This biological response is non-specific because it is the same regardless of the stressor. Its evolution over time has been conceptualised by Hans Selye (1956) in the General Adaptation Syndrome (GAS) which comprises three successive phases. (i) The first phase, known as the alarm phase, corresponds to the activation of all biological mechanisms according to a trend regulation, allowing a rapid response to the stressor. (ii) The second phase of resistance which adjusts the stress response to the intensity of the perceived aggression according to a constant regulation. (iii) When the aggression disappears, a recovery phase dominated by the return of the parasympathetic brake allows a return to homeostasis (eustress).

The "primum movens" of all pathologies is therefore the inability of the individual to adapt his stress response in duration and/or intensity to the course of the phases of the GAS (distress). The perception of not being in control of the situation contributes to the perceived stress and constitutes a well-established risk of distress. It is a risk factor for the emergence of burnout. It induces a biological cost called allostatic cost. Allostasis is a concept that characterizes the process of restoring homeostasis in the presence of a physiological challenge. The term "allostasis" means "achieving stability through change", and refers in part to the process of increasing sympathetic activity and corticotropic axis to promote adaptation and restore homeostasis. Allostasis works well when allostasis systems are initiated when needed and turned off when they are no longer required. Restoring homeostasis involves effective functioning of the parasympathetic system. However, when the allostasis systems remain active, such as during chronic stress, they can cause tissue burnout and accelerate pathophysiological processes.

The perception of uncontrollability depends on the stress situation, the psychological and physiological characteristics of the subject and his or her technical skills in responding to the stressors of the situation. In particular, subjects with a high level of mindfulness are more accepting of uncontrollability and less likely to activate the stress response.

The COVID-19 pandemic situation is a situation characterized by many uncertainties about the individual, family and work environment and the risk of COVID infection. Healthcare workers, like the military, are high-risk occupations that are particularly exposed to these uncertainties in the course of their work and continue to work in an uncertain situation. These professionals are described as a population at risk of occupational/operational burnout that the level of burnout operationalises. This ancillary study in a population of civilian and military non-healthcare workers will complement the study conducted among military health care workers. It will make it possible to isolate the specificity of each profession (civilian or military, healthcare personnel or not) with regard to the risk of burnout in the COVID context.

The objective of this project is to evaluate the impact of the perception of non-control in the operational burnout of experts in their field of practice and to study the psychological and physiological mechanisms mediating the relationship between the subject's characteristics, perceived non-control and burnout.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer personnel i) working at the "Groupement Hospitalier de la Région de Mulhouse Sud Alsace" (GHRMSA) during the COVID-19 crisis OR ii) of the "Groupement Commando Montagne" (GCM) deployed in Mali in June 2020.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to a legal protection measure or unable of giving consent
* Intercurrent pathology with inability to work
* History of psychiatric disorder or cardiac pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of:
  * people who have been working working i) at the "Groupement Hospitalier de la Région de Mulhouse Sud Alsace" (GHRMSA) during the COVID-19 crisis
  * people of the "Groupement Commando Montagne" (GCM) deployed in Mali in June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Professional burnout | 21 days after enrollment (Day 21)
  Professional burnout is measured at D21 by the Burnout Measure Short Version (BMS) questionnaire It is a 10-item questionnaire used to assess burnout regardless of the occupational category.
  Each item is rated from 0 to 6 ("never" to "always"). An average score (sum/10) below 2.4 indicates a very low degree of burnout exposure; a score between 2.5 and 3.4 indicates a low degree of burnout exposure; a score between 3.5 and 4.4 indicates the presence of burnout; a score between 4.5 and 5.4 indicates a high degree of burnout exposure; a score above 5.5 indicates a very high degree of burnout exposure.
Mindfulness level | Day 1
  Mindfulness level is assessed at D0 thanks to the Freiburg Mindfulness Inventory.
  It is a 14 item scale. Each item is rated from 1 to 4 ("almost never" to "almost always"). The total score is between 14 and 56. The mean value in a population of young adults under 36 years of age is 38.5 (+/- 5.1 standard deviation).

SECONDARY OUTCOMES:
Perceived stress level following the emotional stimulation | Day 1
  Perceived stress level is assessed with the Perceived Stress Scale (PSS). It is a 14 item scale. Each item is rated from 0 to 5 ("never" to "very often"). The total score ranges from 0 to 56 with higher scores indicating greater perceived stress.
Parasympathetic flexibility evolution during emotional recall | Day 1
  Parasympathetic flexibility is assessed through dynamic electro-physiological analysis of cardiac and electrodermal conductance recordings.
  Physiological and cognitive reserve of emotional regulation is assessed through the analysis of the spectral power of the 0.1 Hz frequency band at emotional recall.
Sympathetic tone at rest | Day 1
  The activity of the sympathetic tone is assessed by the measurement of the resting state salivary Chromogranin A.
  Physiological and cognitive reserve of emotional regulation is assessed through the analysis of the spectral power of the 0.1 Hz frequency band at emotional recall.
  The activity of the sympathetic tone is assessed by the measurement of the resting salivary Chromogranin A
Corticotropic activation at rest | Day 1
  Corticotropic activation at rest is assessed through the DHEA/cortisol level ratio
Mood disorders (anxiety / depression) | Day 1
  The Hospital Anxiety and Depression Scale (HAD-s32) is used to assess mood disorders in the general non-psychiatric population. It is used to discriminate between anxiety and depression. Scores greater than 11 are indicative of characterized anxiety/depression.
Post-traumatic stress disorder | Day 1
  Post-traumatic disorder is assessed with the PTSD Checklist (PCL-5). It is a 20-item self-administered questionnaire representing Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Post-traumatic stress disorder (PTSD) diagnosis symptoms rated by the subject on a scale from 0 ("not at all") to 4 ("extremely") during the past month. Scores range from 0 to 80. A score greater than of 33 evokes the presence of post-traumatic stress disorder.
Sleep quality | Day 1
  Sleep quality is assesses thanks to the Leeds Sleep Evaluation questionnaire (LEEDS). It consists of ten visual analogue scales assessing four aspects of sleep: (i) quality of falling asleep and degree of drowsiness, (ii) quality of sleep, (iii) quality of wakefulness, and (iv) quality of post-wakefulness and performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Régional de Mulhouse Sud Alsace, Mulhouse, France

IPD SHARING:
Plan to Share IPD: Undecided